CLINICAL TRIAL: NCT05138861
Title: Pharmacokinetic Study to Evaluate the Whole Blood Pharmacokinetics of TP-03 Following Six Week Topical Ocular Administration
Brief Title: A Six Week Pharmacokinetic Study of TP-03 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tarsus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TRS-012
Record Dates: First submitted 2021-07-22; First posted 2021-12-01 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: This is a single-center, open-label, single-arm study.
Masking Description: No masking procedure is required as this is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TP-03 (Lotilaner Ophthalmic Solution), 0.25% (Experimental): TP-03, topical ocular administration in healthy adults. Single and multiple doses for 42 days.
  Interventions: Drug: TP-03 (Lotilaner Ophthalmic Solution), 0.25%

INTERVENTIONS:
Drug: TP-03 (Lotilaner Ophthalmic Solution), 0.25% — A single drop of the ophthalmic solution will be instilled in each eye on the morning of Day 1 and then twice a day (in the morning and in the evening, approximately 12 hours apart) starting on Day 2 for 40 consecutive days (Days 2 to 41). Thereafter, a single drop of the ophthalmic solution will be instilled in each eye on the morning of Day 42, for a total of 82 consecutive doses administered in each eye.

SUMMARY:
Pharmacokinetic Study to Evaluate the Whole Blood Pharmacokinetics of TP-03 Following Six Week Topical Ocular Administration.

DETAILED DESCRIPTION:
This is a single-center, open-label, single-arm study. A single drop of the ophthalmic solution will be instilled in each eye on the morning of Day 1 and then twice a day (in the morning and in the evening, approximately 12 hours apart) starting on Day 2 for 40 consecutive days (Days 2 to 41). Thereafter, a single drop of the ophthalmic solution will be instilled in each eye on the morning of Day 42, for a total of 82 consecutive doses administered in each eye. The doses of Days 1, 2 (morning), 41 (evening), and 42 will be self-administered under supervision of the site staff at the clinical site. All remaining doses will be self-administered at home. Throughout the study, PK blood samples will be collected and safety assessments will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Healthy adult male or female
4. If female, meets one of the following criteria:

   1. Is of childbearing potential and agrees to use an acceptable contraceptive method.

      Or
   2. Male partner has had a vasectomy less than 6 months prior to dosing and the female subject agrees to use an additional acceptable contraceptive method from the first study drug administration until 112 days after the last study drug administration Or
   3. Is of non-childbearing potential, defined as surgically sterile (ie, has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or is in a post-menopausal state (ie, at least 1 year without menses without an alternative medical condition prior to the first study drug administration)
5. Aged at least 18 years
6. Non- or ex-smoker (An ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration)
7. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by an Investigator

Exclusion Criteria:

1. Female who is lactating
2. Female who is pregnant according to the pregnancy test at screening or prior to the first study drug administration
3. Presence or history of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability
4. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
5. Significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
6. Any clinically significant illness in the 28 days prior to the first study drug administration
7. Use of any prescription drugs (with the exception of hormonal contraceptives or hormone replacement therapy) in the 28 days prior to the first study drug administration
8. Use of St. John's wort in the 28 days prior to the first study drug administration
9. History of any ocular surgery or laser within the past 12 months prior to the first study drug administration
10. Have used artificial eyelashes, eyelash extensions or had other cosmetic eyelash or eyelid procedures (e.g., eyeliner tattooing, eyelash tinting, eyelash curling perm, etc.) within 7 days prior to Screening or unwilling to forego their use during the study
11. Presence of clinically significant ocular surface diseases including blepharitis, dry eye, corneal scars, and pterygium, or any ocular abnormalities identified at Screening
12. Presence of acute ocular infection or inflammation at Screening, or required use of eye drops
13. Any history of tuberculosis
14. Positive screening results to HIV Ag/Ab combo, hepatitis B surface antigen or hepatitis C virus tests
15. Intake of an Investigational Product (IP) in the 28 days prior to the first study drug administration
16. Donation of 50 mL or more of blood in the 28 days prior to the first study drug administration
17. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the 56 days prior to the first study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner Cmax at various times
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner Tmax at various times
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner Tlag at various times
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner AUC0-168 at various times
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner AUC0-2880 at various times
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner AUC0-t at various times
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner AUC0-inf at various times
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner CL/F at various times
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner Vz/F at various times
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner eff at various times
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner Thalf at various times
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner λz at various times
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner AUC%extrap at various times
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner MRT0-t at various times
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner Rac at various times
To evaluate the concentration of lotilaner in blood multiple doses of TP-03, 0.25% in whole blood following topical ocular administration in healthy adult subjects for 42 days. | 42 Days
  The primary PK endpoints following single and multiple dose administration will include whole blood PK parameters for lotilaner Ctrough at various times
Incidence of treatment emergent adverse events (TEAEs) | 42 Days
  Safety will be evaluated through the incidence rate of TEAEs
Clinically significant changes from Baseline chemistry laboratory tests | 42 Days
  Evaluate the safety of TP-03 through clinically significant changes from Baseline chemistry laboratory tests
Clinically significant changes from Baseline hematology laboratory tests | 42 Days
  Evaluate the safety of TP-03 through clinically significant changes from Baseline hematology laboratory tests
Clinically significant changes from Baseline physical examinations | 42 Days
  Safety will be evaluated through review of clinically significant changes in physical examinations from Baseline
Clinically significant changes from Baseline electrocardiograms (ECGs) | 42 Days
  Safety will be evaluated through review of clinically significant changes in electrocardiograms from Baseline
Clinically significant changes from Baseline vitals | 42 Days
  Safety will be evaluated through review of clinically significant changes from Baseline vital signs (including temperature [degrees Celsius], pulse rate [beats per minute], respiration rate [breaths per minute], and changes in systolic and diastolic blood pressure [mmHg]) from Baseline
Clinically significant changes from Baseline corrected distance visual acuity | 42 Days
  Safety will be evaluated through review of clinically significant changes in corrected distance visual acuity from Baseline
Clinically significant changes from Baseline non-mydriatic fundus photographs | 42 Days
  Safety will be evaluated through review of clinically significant changes in non-mydriatic fundus photographs from Baseline
Clinically significant changes from Baseline intraocular pressure (IOP) measurement | 42 Days
  Safety will be evaluated through review of clinically significant changes in IOP from Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mark Holdbrook, Study Director — Tarsus Pharmaceuticals
Locations (1):
- Altasciences, Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No